CLINICAL TRIAL: NCT05835843
Title: Study to Assess the Reliability of Psoriasis Area Severity Index Scoring Using Digital-Based Images Compared to In-Person Evaluation
Brief Title: Study to Assess the Reliability of PASI Scoring Using Digital-Based Images
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: INNO-5033
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis; remote assessment; digital photographs
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: ≥0.5 to <5% BSA affected: Approximately 10 subjects with psoriatic plaques covering at least 0.5% but less than 5% of their body surface area
  Interventions: Other: In-Person and Remote Disease Assessment
- Cohort 2: ≥5 to <10% BSA affected: Approximately 10 subjects with psoriatic plaques covering at least 5% but less than 10% of their body surface area
  Interventions: Other: In-Person and Remote Disease Assessment
- Cohort 3: ≥10% BSA affected: Approximately 10 subjects with psoriatic plaques covering at least 10% of their body surface area
  Interventions: Other: In-Person and Remote Disease Assessment

INTERVENTIONS:
Other: In-Person and Remote Disease Assessment — Disease severity will be assessed during the in-person visit and standardized digital photographs of different body regions and/or the full body will be collected for remote evaluations by external dermatologists.

SUMMARY:
This is an open-labeled study to evaluate the reliability of digital photographs for the remote assessment of the disease severity of plaque psoriasis.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the reliability of digital photography for the remote assessment of psoriasis disease severity using the Psoriasis Area and Severity Index (PASI) compared to in-person evaluations. Approximately 30 adult subjects will undergo in-person assessments of the severity of the disease and have digital photographs taken for comparative remote evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 to 75 years, inclusive, at the time of consent.
2. Subject has at least a 6-month history of plaque psoriasis prior to screening visit (information obtained from medical chart or subject's physician, or directly from the subject).
3. Subject has plaque psoriasis covering at least 0.5% his/her total BSA at screening/Day 1 visit.
4. Subject has a PGA score ≥2 at screening/Day 1 visit.

Exclusion Criteria:

1. Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects with at least 0.5% their total BSA affected by plaque psoriasis.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Intraclass Correlation Coefficient (ICC) between Psoriasis Area and Severity Index (PASI) assessed in-person and using digital photographs, all cohorts combined. | Day 1
  The PASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, induration/infiltration, and desquamation (each scored from 0 to 4 separately) for each of 4 body regions, with adjustments for the percentage of BSA involved for each body region and for the proportion of the body region to the whole body.

OTHER OUTCOMES:
Intraclass Correlation Coefficient (ICC) between Physician's Global Assessment (PGA) assessed in-person and using digital photographs, all cohorts combined and by cohort. | Day 1
  The PGA is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity.
Intraclass Correlation Coefficient (ICC) between Body Surface Area (BSA) assessed in-person and using digital photographs, all cohorts combined and by cohort. | Day 1
  The %BSA affected by psoriasis will be evaluated from 1 to 100%.
Intraclass Correlation Coefficient (ICC) between PASI assessed in-person and using digital photographs, by cohort. | Day 1
Intraclass Correlation Coefficient (ICC) of PASI scores assessed using digital photographs by the same assessor. | Day 1
  This outcome measure will assess the variation in PASI scores when evaluated multiple times by the same assessor using digital photographs (intra-rater variability).
Intraclass Correlation Coefficient (ICC) of PASI scores assessed using digital photographs by 2 assessors. | Day 1
  This outcome measure will assess agreement between assessors using digital photographs (inter-rater variability).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research, Montreal, Quebec, Canada